CLINICAL TRIAL: NCT01874548
Title: Magnetic Resonance Study on Metabolism Biomarkers for Cervical Cancer.
Brief Title: MR Metabolic Biomarkers for Cervical Cancer
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Gigin Lin, Department of Radiology, Chang Gung Memorial Hospital
Other Study IDs: 102-0620A3
Record Dates: First submitted 2013-06-06; First posted 2013-06-11 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Autophagy; Cancer metabolism; Cervical cancer; Diffusion weighted imaging; Human papillomavirus; Magnetic resonance spectroscopy.
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tumor tissue will be collected during the operation or biopsy and will be store in liquid nitrogen within 5 minutes removal from body. Standard dual phase tissue extraction will be performed for tumor and cell samples for high resolution MRS analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal cervix: Control group (n=30) comprising surgical candidates with normal cervical tissue will be collected for comparison.
- Cervical cancer: 1. 1st year: 30 surgical candidates with cervical cancer tissue collected during operation.
  2. 2nd year: Enroll another 30 surgical candidates and complete the data regarding clinical MRS/DWI and tissue high resolution MRS. Together with the 30 cancer subjects in part one there will be in total 60 cancer subjects for analysis.
  3. 3rd year: enroll 60 patients primarily treated with CCRT and collect the data using clinical MR and tissue high resolution MRS.

SUMMARY:
The purposes of this study are: (1) to develop magnetic resonance (MR) imaging and spectroscopy as surrogate biomarkers for altered cancer metabolism in cervical cancer; (2) to understand the function of human papillomavirus (HPV) infection and autophagy (a cellular catabolic degradation response to stress) in the metabolic alterations in cervical cancer.

DETAILED DESCRIPTION:
In the first part of this project, we aim to identify the differences in cancer metabolism between normal and cervical cancer. Conventional MR study plus magnetic resonance spectroscopy (MRS) and diffusion weighted imaging (DWI) sequences will be carried out on 30 eligible surgical candidates for pretreatment clinical assessment. Metabolites in cancer tissue will be collected during operation and analyzed using high resolution MRS, and compared with control group comprising 30 patients with normal cervical tissue. The primary endpoint of this part is to identify different MRS profiles between normal and cancer subjects. We will investigate the underlying biological mechanism between these two groups by evaluating status of HPV infection and autophagy. In the second part, we aim to understand cancer metabolism in cervical cancers infected by different types of HPV. We plan to enroll another 30 surgical candidates and complete the data regarding clinical MRS/DWI and tissue high resolution MRS. Together with the 30 cancer subjects in part one there will be in total 60 cancer subjects for analysis. The primary endpoint of this part is to compare MRS profiles from cancer tissue infected with different HPV genotypes, particularly HPV type 16 and HPV type 18. The secondary endpoint is to correlate the tissue MRS profiles with the in vivo MRS/DWI measured by clinical MR scanner. In the third part of this project, we aim to investigate cancer metabolism under combined chemoradiation therapy (CCRT). We plan to enroll 60 patients primarily treated with CCRT and collect the data using clinical MR and tissue high-resolution MRS. Tissue MRS profiles will be correlated with the HPV, E6/E7 and autophagy.

The advance in knowledge of this project is to unwire the complex relationship among cancer metabolism, HPV infection and autophagy in cervical cancer. The clinical impact is the development of MR biomarkers for cancer metabolism and autophagy, both play important roles in the resistance to cancer therapy. The inherited non-invasiveness and non-radiation nature makes MR technique an ideal platform for clinical usage.

ELIGIBILITY:
Inclusion Criteria:

* be able to give informed consent.
* female patients between 20 and 80 years of age.
* biopsy proven newly diagnosed cervical cancer clinical stage International Federation of Gynecology and Obstetrics (FIGO) Ib and above.
* patients must be willing to undergo standard treatment such as surgery or chemo-radiation therapy.

Exclusion Criteria:

* patients who are judged to be noncompliant to treatment or not accessible for follow up.
* patients with contraindications to magnetic resonance imaging (MRI) scanning, such as claustrophobia, cardiac pacemaker, metal implants in field of view, or unable to cooperate for MRI study due to mental status.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in a tertiary referral center.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2013-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
the amounts of metabolites in uterine cervical tissue | up to 8 weeks of magnetic resonance imaging and spectroscopy exam

CONTACTS AND LOCATIONS:
Overall Officials: Gigin Lin, MD, PhD, Principal Investigator — Department of Medical Imaging and Intervention, Chang Gung Memorial Hospital
Locations (1):
- Department of Radiology, Chang Gung Memorial Hospital, Guishan, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin G, Lai CH, Tsai SY, Lin YC, Huang YT, Wu RC, Yang LY, Lu HY, Chao A, Wang CC, Ng KK, Ng SH, Chou HH, Yen TC, Hung JH. 1 H MR spectroscopy in cervical carcinoma using external phase array body coil at 3.0 Tesla: Prediction of poor prognostic human papillomavirus genotypes. J Magn Reson Imaging. 2017 Mar;45(3):899-907. doi: 10.1002/jmri.25386. Epub 2016 Jul 19. PMID 27434095
- See also: 1 H MR spectroscopy in cervical carcinoma using external phase array body coil at 3.0 Tesla: Prediction of poor prognostic human papillomavirus genotypes. — http://www.ncbi.nlm.nih.gov/pubmed/27434095